CLINICAL TRIAL: NCT02182232
Title: A Phase I Open Label Dose Escalation Study of Continuous Oral Treatment With BIBF 1120 Together With Paclitaxel and Carboplatin in Patients With Advanced Stage Non-small-cell Lung Cancer
Brief Title: A Dose Escalation Study of BIBF 1120 Together With Paclitaxel and Carboplatin in Patients With Advanced Stage Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.5
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — nintedanib; Paclitaxel; Carboplatin

ARMS (2):
- BIBF 1120 with paclitaxel and carboplatin (Experimental)
  Interventions: Drug: BIBF 1120; Drug: Paclitaxel; Drug: Carboplatin
- BIBF 1120 monotherapy (Experimental)
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: BIBF 1120
  Arms: BIBF 1120 with paclitaxel and carboplatin
Drug: Paclitaxel
  Arms: BIBF 1120 with paclitaxel and carboplatin
Drug: Carboplatin

SUMMARY:
The primary objectives of this trial were to determine the MTD of BIBF 1120 in combination with carboplatin and paclitaxel, pharmacokinetics and objective response of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with histologically or cytologically confirmed Stage IIIB (including pleural effusion), IV or recurrent NSCLC
2. Bi-dimensionally measurable disease by one or more techniques (CT, MRI, X-ray)
3. Age 18 years or older
4. Life expectancy of at least three (3) months
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
6. Written informed consent that is consistent with ICH-GCP guidelines

Exclusion Criteria:

1. Prior treatment for NSCLC including chemotherapy, biologic response modifier therapy, or any investigational drug
2. Participation in another clinical study within the past four weeks before start of therapy or concomitantly with this study
3. Active brain metastases (stable for <28 days, symptomatic, or requiring concurrent steroids or antiepileptic therapy)
4. Centrally located tumors with radiologic evidence (CT or MRI) of local invasion of major blood vessels
5. Cavitary or necrotic tumors
6. Sanguinous pleural effusion due to disease or pericardial effusion suspicious for disease
7. Radiotherapy to an area of measurable disease (unless disease progression had been documented following completion of therapy)
8. Radiotherapy within 4 weeks preceding Day 0
9. Other active malignancy diagnosed within the past 3 years (other than non-melanomatous skin cancer)
10. Gastrointestinal abnormalities that would interfere with intake or absorption of the study drug, such as a requirement for intravenous alimentation, prior surgical procedures affecting absorption, treatment for peptic ulcer disease within the last 6 months, active gastrointestinal bleeding unrelated to cancer (as evidenced by either hematemesis, hematochezia, or melena in the past 3 months and without endoscopic documented resolution), or malabsorption syndromes
11. Significant cardiovascular disease (i.e., uncontrolled hypertension, myocardial infarction within 6 months, unstable angina, serious cardiac arrhythmia, ≥NYHA Grade 2 congestive heart failure)
12. History of hemorrhagic or thrombotic event (including transient ischemic attacks) in the past 12 months
13. Clinically significant hemoptysis (1 teaspoon or more) in the past 3 months
14. Concurrent therapeutic anticoagulation (except heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except chronic low-dose daily aspirin <325 mg)
15. Known hypersensitivity to paclitaxel, carboplatin, or any of their excipients including Cremophor® (polyoxyethylated castor oil)
16. Absolute neutrophil count (ANC) ≤1,500/μl, platelet count ≤100,000/μl, or hemoglobin <9 gm/dL
17. Total bilirubin >1.5 mg/dL (26 μmol/L, SI Unit equivalent), alanine amino transferase (ALT) and/or aspartate amino transferase (AST) ≥1.5 X ULN,
18. Serum creatinine >1.5 mg/dL (>132 μmol/L, SI Unit equivalent)
19. Persistent hematuria or proteinuria (more than trace)
20. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
21. Pregnancy or breastfeeding
22. Known or suspected active alcohol or drug abuse
23. Patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Incidence and intensity of adverse events according to Common Terminology Criteria for Adverse Events (version 3.0) associated with increasing doses of BIBF 1120 | up to day 126
Maximum tolerated dose (MTD) of BIBF 1120 in combination with carboplatin and paclitaxel | up to day 21

SECONDARY OUTCOMES:
Pre-dose plasma concentration (Cpre) | up to day 42
Objective tumor response according to response evaluation criteria in solid tumors (RECIST) | up to 12 months
Time from best response to onset of tumor progression | Up to 12 months
Time from start of treatment to time of documented tumor progression | Up to 12 months
area under the curve (AUC) from 0 to 12 hours (AUC0-12) | up to day 42
AUC from 0 to the last quantifiable drug concentration (AUC0-tz) | up to day 42
Maximum plasma concentration (Cmax) | up to day 42
Time to maximum plasma concentration (tmax) | up to day 42
Rate constant (λz) for BIBF 1120 | up to day 42
AUC from 0 to 24 hours (AUC0-24) for paclitaxel | up to day 42
AUC from 0 extrapolated to 48 hours (AUC0-48) for paclitaxel | up to day 42
AUC from 0 extrapolated to infinity (AUC0-∞) | up to day 42
Percentage of AUC0-∞ that is obtained by extrapolation (% AUCtz-∞) | up to day 42
Terminal half-life (t1/2) | up to day 42
Mean residence time after intravenous administration (MRTiv) for paclitaxel and carboplatin | up to day 42
Total Clearance (CL/F) | up to day 42
Volume of distribution during the terminal phase (Vz) | up to day 42
AUC from 0 to 24 hours (AUC0-24) for carboplatin | Day 1 and 22 in the treatment time
Plasma concentration 21 hours after start of infusion (C21) for carboplatin | up to day 42
Plasma concentration 24 hours after start of infusion (C24) for paclitaxel | up to day 42